CLINICAL TRIAL: NCT01475721
Title: SAS115359, a Safety and Efficacy Study of Inhaled Fluticasone Propionate/Salmeterol Combination Versus Inhaled Fluticasone Propionate in the Treatment of Adolescent and Adult Subjects With Asthma
Brief Title: SAS115359: A 6-month Study to Assess the Safety and Benefit of Inhaled Fluticasone Propionate/Salmeterol Combination Compared With Inhaled Fluticasone Propionate in the Treatment of Adolescents and Adults (12 Years of Age and Older) With Asthma.
Acronym: AUSTRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 115359
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Asthma
Keywords: ADVAIR; Asthma; safety; FLOVENT
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- ADVAIR 100/50mcg (Experimental): experimental drug
  Interventions: Drug: ADVAIR 100/50mcg
- ADVAIR 250/50mcg (Experimental): experimental drug
  Interventions: Drug: ADVAIR 250/50mcg
- ADVAIR 500/50mcg (Experimental): experimental drug
  Interventions: Drug: ADVAIR 500/50mcg
- FLOVENT 100mcg (Active Comparator): active comparator
  Interventions: Drug: FLOVENT 100mcg
- FLOVENT 250mcg (Active Comparator): active comparator
  Interventions: Drug: FLOVENT 250mcg
- FLOVENT 500mcg (Active Comparator): active comparator
  Interventions: Drug: FLOVENT 500mcg

INTERVENTIONS:
Drug: ADVAIR 100/50mcg — fluticasone propionate/salmeterol combination (100/50mcg) twice daily (AM and PM) for 6 months
  Other Names: FSC 100/50
  Arms: ADVAIR 100/50mcg
Drug: ADVAIR 250/50mcg — fluticasone propionate/salmeterol combination (250/50mcg) twice daily (AM and PM) for 6 months
  Other Names: FSC 250/50
  Arms: ADVAIR 250/50mcg
Drug: ADVAIR 500/50mcg — fluticasone propionate/salmeterol combination (500/50mcg) twice daily (AM and PM) for 6 months
  Other Names: FSC 500/50
  Arms: ADVAIR 500/50mcg
Drug: FLOVENT 100mcg — fluticasone propionate (100) twice daily (AM and PM) for 6 months
  Other Names: FP 100
  Arms: FLOVENT 100mcg
Drug: FLOVENT 250mcg — fluticasone propionate (250mcg) twice daily (AM and PM) for 6 months
  Other Names: FP 250
  Arms: FLOVENT 250mcg
Drug: FLOVENT 500mcg — fluticasone propionate (500mcg) twice daily (AM and PM) for 6 months
  Other Names: FP 500
  Arms: FLOVENT 500mcg

SUMMARY:
The purpose of this study is to assess whether the risk of serious asthma-related events (asthma-related hospitalizations, endotracheal intubations, and deaths) in adolescents and adults (12 years of age and older) taking inhaled fluticasone propionate/salmeterol combination is the same as those taking inhaled fluticasone propionate alone.

ADVAIR™ and FLOVENT™ are trademarks of the GlaxoSmithKline Group of Companies.

DETAILED DESCRIPTION:
Progress of Enrollment, Updated Annually: This study has been completed and the final clinical study report was submitted to the FDA in January of 2016. This is the final update, as this study is complete.

ELIGIBILITY:
Inclusion Criteria:

* Provided consent to participate in the study
* Male or female, 12 years of age and older
* Clinical diagnosis of asthma for at least 1 year prior to the randomization
* Clinic PEF of greater than or equal to 50% of predicted normal value
* Subject must be appropriately using one of the treatments for asthma listed in the protocol
* Subject must be able to complete the asthma control questionnaire, daily questions about asthma, and use a DISKUS inhaler
* Subject must have history of at least 1 asthma exacerbation including one of the following in the year prior to randomization:
* requiring treatment with systemic corticosteroids
* an asthma-related hospitalization

Exclusion Criteria:

* History of life threatening asthma defined for this protocol as asthma episode that required intubation and/or was associated with hypercapnea requiring non-invasive ventilatory support
* Concurrent respiratory disease other than asthma
* Current evidence of, or ever been told by a physician that they have chronic bronchitis, emphysema, or chronic obstructive pulmonary disease.
* Exercise induced asthma (as the only asthma-related diagnosis) not requiring daily asthma control medicine
* Presence of a bacterial or viral respiratory infection that is not resolved at randomization
* An asthma exacerbation requiring systemic corticosteriods within 4 weeks of randomization or more than 4 separate exacerbations in the 12 months preceding randomization
* More than 2 hospitalizations for treatment of asthma in the 12 months preceding randomization
* Subject must not meet unstable asthma severity criteria as listed in the protocol
* Potent cytochrome P450 3A4 (CYP3A4) inhibitors within the last 4 weeks (e.g., ritonavir, ketoconazole, itraconzole)
* Pregnancy, breast-feeding or planned pregnancy during the study
* A Child in Care (CiC) is a child who has been placed under the control or protection of an agency, organisation, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11751 (Actual)
Dates: Start 2011-11-18 (Actual); Primary Completion 2015-06-23 (Actual); Study Completion 2015-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (617):
- United States (276):
  - GSK Investigational Site, Athens, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Florence, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Pell City, Alabama
  - GSK Investigational Site, Scottsboro, Alabama
  - GSK Investigational Site, Toney, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Flagstaff, Arizona
  - GSK Investigational Site, Goodyear, Arizona
  - GSK Investigational Site, Green Valley, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Sierra Vista, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Dinuba, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Granada Hills, California
  - GSK Investigational Site, Harbor City, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, Lomita, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Napa, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Pismo Beach, California
  - GSK Investigational Site, Pomona, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Gabriel, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, San Marcos, California
  - GSK Investigational Site, San Marino, California
  - GSK Investigational Site, San Ramon, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Ventura, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, West Sacramento, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Thornton, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Danbury, Connecticut
  - GSK Investigational Site, Milford, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Destin, Florida
  - GSK Investigational Site, Doral, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Jupiter, Florida
  - GSK Investigational Site, Maitland, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Trinity, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Wellington, Florida
  - GSK Investigational Site, Zephyrhills, Florida
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Lilburn, Georgia
  - GSK Investigational Site, Rincon, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Tucker, Georgia
  - GSK Investigational Site, Champaign, Illinois
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, Glen Ellyn, Illinois
  - GSK Investigational Site, Glenview, Illinois
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Oak Lawn, Illinois
  - GSK Investigational Site, Oak Park, Illinois
  - GSK Investigational Site, Shiloh, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Brownsburg, Indiana
  - GSK Investigational Site, Crown Point, Indiana
  - GSK Investigational Site, Franklin, Indiana
  - GSK Investigational Site, Greenfield, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Muncie, Indiana
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Hutchinson, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Hazard, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Alexandria, Louisiana
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Portland, Maine
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Hollywood, Maryland
  - GSK Investigational Site, Largo, Maryland
  - GSK Investigational Site, Silver Spring, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Wheaton, Maryland
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Hyannis, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Buckley, Michigan
  - GSK Investigational Site, Chelsea, Michigan
  - GSK Investigational Site, Chesterfield, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Fenton, Michigan
  - GSK Investigational Site, Interlochen, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Niles, Michigan
  - GSK Investigational Site, Novi, Michigan
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Port Gibson, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Atco, New Jersey
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, Freehold, New Jersey
  - GSK Investigational Site, Lumberton, New Jersey
  - GSK Investigational Site, Marlton, New Jersey
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Ridgewood, New Jersey
  - GSK Investigational Site, Trenton, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Corning, New York
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, New Windsor, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Newburgh, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Utica, New York
  - GSK Investigational Site, Westfield, New York
  - GSK Investigational Site, Asheboro, North Carolina
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Calabash, North Carolina
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Clyde, North Carolina
  - GSK Investigational Site, Lexington, North Carolina
  - GSK Investigational Site, Morganton, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Centerville, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Groveport, Ohio
  - GSK Investigational Site, Marion, Ohio
  - GSK Investigational Site, Middleburg Heights, Ohio
  - GSK Investigational Site, Shaker Heights, Ohio
  - GSK Investigational Site, Springfield, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Wheeling, Ohio
  - GSK Investigational Site, Youngstown, Ohio
  - GSK Investigational Site, Zanesville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Belle Vernon, Pennsylvania
  - GSK Investigational Site, Bensalem, Pennsylvania
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Downingtown, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Holland, Pennsylvania
  - GSK Investigational Site, Huntingdon Valley, Pennsylvania
  - GSK Investigational Site, Jenkintown, Pennsylvania
  - GSK Investigational Site, Lansdale, Pennsylvania
  - GSK Investigational Site, Latrobe, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Scottdale, Pennsylvania
  - GSK Investigational Site, Shippensburg, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, East Greenwich, Rhode Island
  - GSK Investigational Site, Johnston, Rhode Island
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Florence, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Greenwood, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Dakota Dunes, South Dakota
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, McKenzie, Tennessee
  - GSK Investigational Site, Shelbyville, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Duncanville, Texas
  - GSK Investigational Site, Gun Barrel City, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, Killeen, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Lufkin, Texas
  - GSK Investigational Site, McKinney, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Clinton, Utah
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Midvale, Utah
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Falls Church, Vermont
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Midlothian, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Suffolk, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Port Orchard, Washington
  - GSK Investigational Site, Puyallup, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Morgantown, West Virginia
  - GSK Investigational Site, Madison, Wisconsin
- Argentina (12):
  - GSK Investigational Site, Derqui, Pilar, Buenos Aires
  - GSK Investigational Site, Nueve de Julio, Buenos Aires
  - GSK Investigational Site, San Martín, Buenos Aires
  - GSK Investigational Site, Concepción del Uruguay, Entre Ríos Province
  - GSK Investigational Site, Paraná, Entre Ríos Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, Lanús
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Rosario
- Australia (10):
  - GSK Investigational Site, Broadmeadow, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Redcliffe, Queensland
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Subiaco, Western Australia
  - GSK Investigational Site, Parkville
- Austria (4):
  - GSK Investigational Site, Feldkirch
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
  - GSK Investigational Site, Wels
- Belgium (5):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Jambes
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Montigny-le-Tilleul
  - GSK Investigational Site, Natoye
- Bulgaria (9):
  - GSK Investigational Site, Blagoevgrad
  - GSK Investigational Site, Pazardzhik
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sliven
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Troyan Municipality
  - GSK Investigational Site, Varna
  - GSK Investigational Site, Veliko Tarnovo
  - GSK Investigational Site, Vidin
- Canada (12):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Fort Erie, Ontario
  - GSK Investigational Site, Grimsby, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
- Chile (5):
  - GSK Investigational Site, Temuco, Región de La Araucania
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Valdivia
  - GSK Investigational Site, Viña del Mar
- Colombia (2):
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Bucaramanga
- Croatia (4):
  - GSK Investigational Site, Čakovec
  - GSK Investigational Site, Senj
  - GSK Investigational Site, Zadar
  - GSK Investigational Site, Zagreb
- Czechia (8):
  - GSK Investigational Site, Havlíčkův Brod
  - GSK Investigational Site, Hlučín
  - GSK Investigational Site, Jaroměř
  - GSK Investigational Site, Kyjov
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Svitavy
  - GSK Investigational Site, Třemošná
- Denmark (2):
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Rosklide
- Germany (65):
  - GSK Investigational Site, Bruchsal, Baden-Wurttemberg
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Bad Woerrishofen, Bavaria
  - GSK Investigational Site, Feldkirchen, Bavaria
  - GSK Investigational Site, Fürth, Bavaria
  - GSK Investigational Site, Gars Am Inn, Bavaria
  - GSK Investigational Site, Georgensgmünd, Bavaria
  - GSK Investigational Site, Großheirath, Bavaria
  - GSK Investigational Site, Höchstadt an der Aisch, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Neuötting, Bavaria
  - GSK Investigational Site, Vilshofen, Bavaria
  - GSK Investigational Site, Weißenhorn, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Rathenow, Brandenburg
  - GSK Investigational Site, Bad Arolsen, Hesse
  - GSK Investigational Site, Bensheim, Hesse
  - GSK Investigational Site, Frankenberg, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Lahnau, Hesse
  - GSK Investigational Site, Offenbach, Hesse
  - GSK Investigational Site, Rodgau, Hesse
  - GSK Investigational Site, Rüsselsheim am Main, Hesse
  - GSK Investigational Site, Schwalmstadt, Hesse
  - GSK Investigational Site, Bad Pyrmont, Lower Saxony
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Wolfsburg, Lower Saxony
  - GSK Investigational Site, Bad Lippspringe, North Rhine-Westphalia
  - GSK Investigational Site, Beckum, North Rhine-Westphalia
  - GSK Investigational Site, Bergisch Gladbach, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Engelskirchen, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Hagen, North Rhine-Westphalia
  - GSK Investigational Site, Herne, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Ratingen, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Telgte, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Wuppertal, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Raubach, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Dillingen, Saarland
  - GSK Investigational Site, Saarbrücken, Saarland
  - GSK Investigational Site, Auerbach, Saxony
  - GSK Investigational Site, Böhlen, Saxony
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Meissen, Saxony
  - GSK Investigational Site, Teuchern, Saxony-Anhalt
  - GSK Investigational Site, Zerbst, Saxony-Anhalt
  - GSK Investigational Site, Klappholz, Schleswig-Holstein
  - GSK Investigational Site, Reinfeld, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hungary (11):
  - GSK Investigational Site, Baja
  - GSK Investigational Site, Balassagyarmat
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Kaposvár
  - GSK Investigational Site, Komló
  - GSK Investigational Site, Mosonmagyaróvár
  - GSK Investigational Site, Nagykanizsa
  - GSK Investigational Site, Ráckeve
  - GSK Investigational Site, Siófok
  - GSK Investigational Site, Szolnok
- Indonesia (8):
  - GSK Investigational Site, Denpasar
  - GSK Investigational Site, Depok Timur
  - GSK Investigational Site, Jakarta
  - GSK Investigational Site, Malang
  - GSK Investigational Site, Medan
  - GSK Investigational Site, Palembang
  - GSK Investigational Site, Semarang
  - GSK Investigational Site, Surakarta
- Italy (15):
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Arenzano, Liguria
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Messina
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Monza
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Sesto San Giovanni
- Latvia (3):
  - GSK Investigational Site, Kuldīga
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Tukums
- Lithuania (5):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Šiauliai
  - GSK Investigational Site, Utena
  - GSK Investigational Site, Vilnius
- Malaysia (5):
  - GSK Investigational Site, Alor Star
  - GSK Investigational Site, Kota Bharu
  - GSK Investigational Site, Kuala Pilah
  - GSK Investigational Site, Kuala Selangor
  - GSK Investigational Site, Sungai Buloh
- Mexico (6):
  - GSK Investigational Site, Aguascalientes, Ags, Aguascalientes
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Huixquilucan
  - GSK Investigational Site, Monterrey
  - GSK Investigational Site, Zapopan
- Peru (2):
  - GSK Investigational Site, Lima
  - GSK Investigational Site, San Borja, Lima
- Philippines (6):
  - GSK Investigational Site, Dasmariñas, Cavite
  - GSK Investigational Site, Davao City
  - GSK Investigational Site, Las Piñas
  - GSK Investigational Site, Los Baños
  - GSK Investigational Site, Pulilan
  - GSK Investigational Site, Quezon City
- Poland (30):
  - GSK Investigational Site, Bielsko-Biala
  - GSK Investigational Site, Brzesko
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Bystra
  - GSK Investigational Site, Cieszyn
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Głuchołazy
  - GSK Investigational Site, Jelenia Góra
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Libiąż
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lubin
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Radomsko
  - GSK Investigational Site, Ruda Śląska
  - GSK Investigational Site, Rudka
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Sandomierz
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wodzisław Śląski
  - GSK Investigational Site, Wołomin
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zabrze
  - GSK Investigational Site, Zgierz
- Romania (3):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Sibiu
- Russia (17):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Kirov
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Orenburg
  - GSK Investigational Site, Pyatigorsk
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Veliky Novgorod
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
- GSK Investigational Site, Belgrade, Serbia
- Slovakia (6):
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Kráľovský Chlmec
  - GSK Investigational Site, Levice
  - GSK Investigational Site, Martin
  - GSK Investigational Site, Štúrovo
  - GSK Investigational Site, Trnava
- South Africa (18):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Cape Town, Gauteng
  - GSK Investigational Site, Eloffsdal, Gauteng
  - GSK Investigational Site, Krugersdorp, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Benoni
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Claremont
  - GSK Investigational Site, Die Wilgers
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Gatesville
  - GSK Investigational Site, Middelburg
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Soweto
  - GSK Investigational Site, Thabazimbi
  - GSK Investigational Site, Welkom
- South Korea (6):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Chuncheon
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (22):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Basurto/Bilbao
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Canet de Mar - Barcelona
  - GSK Investigational Site, Elche
  - GSK Investigational Site, Illescas-Toledo
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Sagunto/Valencia
  - GSK Investigational Site, Sant Boi de Llobregat
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Tarrasa, Barcelona
  - GSK Investigational Site, Torrelavega
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Vic (Barcelona)
- Taiwan (5):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Keelung
  - GSK Investigational Site, Koahsiung
  - GSK Investigational Site, Putzu
  - GSK Investigational Site, Taipei
- Ukraine (18):
  - GSK Investigational Site, Cherkassy
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kryvyi Rih
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Sumy
  - GSK Investigational Site, Ternopil
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhzhia
  - GSK Investigational Site, Zaporizhzhya
  - GSK Investigational Site, Zhytomyr
- United Kingdom (16):
  - GSK Investigational Site, Bedford, Bedfordshire
  - GSK Investigational Site, Cardiff, Glamorgan
  - GSK Investigational Site, Manchester, Greater Manchester
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Bath, Somerset
  - GSK Investigational Site, Brighton, Sussex East
  - GSK Investigational Site, Barry
  - GSK Investigational Site, Bexhill-on-Sea
  - GSK Investigational Site, Chertsey, Surrey
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Kent
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, London
  - GSK Investigational Site, Merseyside
  - GSK Investigational Site, Penzance
  - GSK Investigational Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Busse W, Stempel D, Aggarwal B, Boucot I, Forth R, Raphiou I, Rabe KF, Reddel HK. Insights from the AUSTRI study on reliever use before and after asthma exacerbations. J Allergy Clin Immunol Pract. 2022 Jul;10(7):1916-1918.e2. doi: 10.1016/j.jaip.2022.03.029. Epub 2022 Apr 9. No abstract available. PMID 35413473
- [Derived] Stempel DA, Raphiou IH, Kral KM, Yeakey AM, Emmett AH, Prazma CM, Buaron KS, Pascoe SJ; AUSTRI Investigators. Serious Asthma Events with Fluticasone plus Salmeterol versus Fluticasone Alone. N Engl J Med. 2016 May 12;374(19):1822-30. doi: 10.1056/NEJMoa1511049. Epub 2016 Mar 6. PMID 26949137
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 115359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study duration was 29 weeks, comprised of a randomization visit followed by a treatment period of 26 weeks and a 1 week follow-up phone call. Participants were assessed for eligibility at screening up to 15 days prior to randomization.
Pre-assignment Details: Eligible adolescent and adult participants with asthma were stratified based on current asthma medication and a Asthma Control Questionnaire (ACQ-6) score and randomized 1:1 to double-blind study treatment. A total of 11751 were enrolled; however, 72 were randomized but did not receive study treatment.
Groups:
- Fluticasone Propionate/Salmeterol Combination (FSC): Participants received one of following treatments: FSC 100/50 microgram (µg) or FSC 250/50 µg or FSC 500/50 µg as one inhalation twice daily (BID) via Dry powder inhaler (DPI) for 26 weeks. Rescue medication (albuterol/salbutamol) via metered dose inhaler (MDI) was permitted during study treatment. Participants were instructed to stop using their current asthma medication.
- Fluticasone Propionate (FP): Participants received one of following treatments: FP 100 µg or FP 250 µg or FP 500 µg as one inhalation (BID) via (DPI) for 26 weeks. Rescue medication (albuterol/salbutamol) via metered dose inhaler (MDI) was permitted during study treatment. Participants were instructed to stop using their current asthma medication.
Period: Overall Study
Arm/Group | Fluticasone Propionate/Salmeterol Combination (FSC) | Fluticasone Propionate (FP)
Started | 5834 | 5845
Completed | 5823 | 5831
Not Completed | 11 | 14
Not completed — Death | 3 | 6
Not completed — Withdrawal by Subject | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate/Salmeterol Combination (FSC) | Fluticasone Propionate (FP) | Total
Number analyzed (Participants) | 5834 | 5845 | 11679
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (17.45) | 43.4 (17.28) | 43.4 (17.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3851 | 3898 | 7749
  Male | 1983 | 1947 | 3930
Race/Ethnicity, Customized [Number; unit: Participants]
  Missing | 3 | 3 | 6
  African American/African Heritage | 870 | 856 | 1726
  American Indian/Alaska native | 109 | 116 | 225
  Asian-Central/South Asian Heritage | 36 | 45 | 81
  Asian-East Asian Heritage | 94 | 88 | 182
  Japanese Heritage | 4 | 3 | 7
  Asian-South East Asian Heritage | 234 | 224 | 458
  Native Hawaiian or other Pacific Islander | 8 | 10 | 18
  White-Arabic/North African Heritage | 22 | 21 | 43
  White-White/Caucasian/European Heritage | 4352 | 4388 | 8740
  Multiple | 102 | 91 | 193

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing an Event in the Composite Safety Endpoint of Serious Asthma Outcomes ( Asthma-related Hospitalization, Asthma-related Endotracheal Intubation, or Asthma-related Death)
Description: Composite endpoint was defined as clinically relevant endpoint that is constructed from combinations of other clinically relevant endpoints of serious asthma outcomes (i.e., asthma-related hospitalization, asthma-related endotracheal intubation, or asthma-related death). Hospitalization was defined as an inpatient stay or a ≥24-hour stay in an observation area in an emergency department or other equivalent facility. Probability of having event was summarized with Kaplan-Meier estimates.Hazard ratio, confidence interval, and p-value are from a stratified Cox proportional hazard model, using randomization stratum as the stratification factor. The 95% CI provided in the table is actually the 95.
Time Frame: From Day 1 up to 26 weeks
Population: Intent to treat (ITT) Population comprised of all participants randomized to study drug and who took study drug.
Measure: Number; unit: Participants
Arm/Group | Fluticasone Propionate/Salmeterol Combination (FSC) | Fluticasone Propionate (FP)
Number analyzed (Participants) | 5834 | 5845
Participants | 34 | 33
Statistical Analysis 1: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); Test type: Non-Inferiority or Equivalence — The non-inferiority comparison is statistically significant if the upper bound of the two-sided 95% CI falls below 2, the non-inferiority margin, and the non-inferiority test one-sided p-value <0.025; p = 0.003, Regression, Cox; Hazard Ratio (HR) = 1.029, 95% CI 2-sided [0.638 to 1.662]

2. Primary Outcome: Number of Participants Experiencing at Least One Asthma Exacerbation
Description: An asthma exacerbation is defined as a deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least three days or an inpatient hospitalization or emergency department visit due to asthma that required systemic corticosteroids.
Time Frame: From Day 1 up to 26 weeks
Population: Modified intent to treat (mITT) Population comprised of participants included in the ITT population that correspond to each participant's period of exposure to study drug plus seven days after the last date of study drug treatment.
Measure: Number; unit: Participants
Arm/Group | Fluticasone Propionate/Salmeterol Combination (FSC) | Fluticasone Propionate (FP)
Number analyzed (Participants) | 5834 | 5845
Participants | 480 | 597
Statistical Analysis 1: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); The hazard ratio computed is essentially the relative risk of having the event in the treatment group relative to the control group, adjusted for time to the event; Test type: Superiority or Other; p = 0.203, Regression, Cox; Hazard Ratio (HR) = 0.834, 95% CI 2-sided [0.630 to 1.103] — Analysis of time to first exacerbation in efficacy subgroup: Subjects not well-controlled on prior ICS or non-LABA therapy
Statistical Analysis 2: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.188, Regression, Cox; Hazard Ratio (HR) = 0.839, 95% CI 2-sided [0.645 to 1.090] — Analysis of time to first exacerbation in efficacy subgroup: Subjects not well-controlled on prior ICS+LABA therapy
Statistical Analysis 3: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 0.764, 95% CI 2-sided [0.645 to 0.905] — Analysis of time to first exacerbation in efficacy subgroup: Subjects controlled on prior ICS+LABA therapy
Statistical Analysis 4: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.071, Regression, Cox; Hazard Ratio (HR) = 0.682, 95% CI 2-sided [0.451 to 1.034] — Analysis of time to first exacerbation in efficacy subgroup: Subjects controlled on prior ICS therapy
Statistical Analysis 5: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.373, Regression, Cox; Hazard Ratio (HR) = 0.878, 95% CI 2-sided [0.659 to 1.170] — Analysis of number of asthma exacerbations in efficacy subgroup: Subjects not well-controlled on prior ICS or non-LABA therapy
Statistical Analysis 6: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.271, Regression, Cox; Hazard Ratio (HR) = 0.864, 95% CI 2-sided [0.665 to 1.122] — Analysis of number of asthma exacerbations in efficacy subgroup: Subjects not well-controlled on prior ICS+LABA therapy
Statistical Analysis 7: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 0.755, 95% CI 2-sided [0.637 to 0.895] — Analysis of number of asthma exacerbations in efficacy subgroup: Subjects controlled on prior ICS+LABA therapy
Statistical Analysis 8: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.075, Regression, Cox; Hazard Ratio (HR) = 0.687, 95% CI 2-sided [0.454 to 1.040] — Analysis of number of asthma exacerbations in efficacy subgroup: Subjects controlled on prior ICS therapy

3. Secondary Outcome: Number of Participants Experiencing at Least One Asthma Related Hospitalization , Endotracheal Intubation and Death
Description: Hospitalization was defined as an inpatient stay or a ≥24-hour stay in an observation area in an emergency department or other equivalent facility.
Time Frame: From Day 1 up to 26 weeks
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Fluticasone Propionate/Salmeterol Combination (FSC) | Fluticasone Propionate (FP)
Number analyzed (Participants) | 5834 | 5845
Participants
  Hospitalization | 34 | 33
  Endotracheal intubation | 0 | 2
  Death | 0 | 0

4. Secondary Outcome: Number of Participant Withdrawals From Study Treatment Due to Asthma Exacerbation
Description: as for outcome 2
Time Frame: From Day 1 up to 26 weeks
Population: mITT Population
Measure: Number; unit: Participants
Arm/Group | Fluticasone Propionate/Salmeterol Combination (FSC) | Fluticasone Propionate (FP)
Number analyzed (Participants) | 5834 | 5845
Participants | 66 | 84
Statistical Analysis 1: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); Test type: Superiority or Other; p = 0.123, Regression, Cox; Hazard Ratio (HR) = 0.776, 95% CI 2-sided [0.562 to 1.071]

5. Secondary Outcome: Mean Rescue Medication (Albuterol/Salbutamol) Use as Puffs Per 24 Hours
Description: Rescue medication included albuterol/salbutamol used to treat acute asthma were reported as puffs per 24 hours over a period of 6 months.
Time Frame: From Day 1 up to 26 weeks
Population: mITT Population. Only those participants available at specified timepoint were analysed.
Measure: Mean (Standard Error); unit: Number of Puffs
Arm/Group | Fluticasone Propionate/Salmeterol Combination (FSC) | Fluticasone Propionate (FP)
Number analyzed (Participants) | 5677 | 5673
Number of Puffs | 0.90 (0.018) | 1.09 (0.020)
Statistical Analysis 1: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); Test type: Superiority or Other; p < 0.001, Regression, Cox; Mean Difference (Final Values) = -0.263, 95% CI 2-sided [-0.385 to -0.141] — Efficacy subgroup: Subjects not well-controlled on prior ICS or non-LABA therapy
Statistical Analysis 2: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); Test type: Superiority or Other; p = 0.003, Regression, Cox; Mean Difference (Final Values) = -0.222, 95% CI 2-sided [-0.369 to -0.076] — Efficacy subgroup: Subjects not well-controlled on prior ICS+LABA therapy
Statistical Analysis 3: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); Test type: Superiority or Other; p < 0.001, Regression, Cox; Mean Difference (Final Values) = -0.172, 95% CI 2-sided [-0.238 to -0.106] — Efficacy subgroup: Subjects controlled on prior ICS+LABA therapy
Statistical Analysis 4: Comparison: Fluticasone Propionate/Salmeterol Combination (FSC) vs Fluticasone Propionate (FP); Test type: Superiority or Other; p = 0.251, Regression, Cox; Mean Difference (Final Values) = -0.080, 95% CI 2-sided [-0.216 to 0.056] — Efficacy subgroup: Subjects controlled on prior ICS therapy

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious events (AEs) were collected from post-randomization, throughout the treatment period of 26 weeks up to a 1-week follow-up phone call (27 Weeks).
Description: All SAEs are presented and Non-serious AEs were collected from the members of mITT population up until the participants' withdrawal from study treatment, only non-serious AEs that lead to withdrawal of study treatment were collected
Arm/Group | Fluticasone Propionate/Salmeterol Combination (FSC) | Fluticasone Propionate (FP)
Serious Adverse Events (participants affected / at risk) | 134/5834 | 125/5845
Other Adverse Events (participants affected / at risk) | 46/5834 | 75/5845
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluticasone Propionate/Salmeterol Combination (FSC) (N=5834) | Fluticasone Propionate (FP) (N=5845)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1)
Hereditary angioedema (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 2 (2) | 4 (5)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (3)
Allergic granulomatous angiitis (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (3)
Pyelonephritis (Infections and infestations) | 3 (3) | 0 (0)
Dengue fever (Infections and infestations) | 2 (2) | 0 (0)
Typhoid fever (Infections and infestations) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8) | 8 (9)
Salpingo-oophoritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Coagulation time prolonged (Investigations) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (2) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Spinal subdural haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 3 (3)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Stress (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Bulimia nervosa (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Somnambulism (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Fallopian tube cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine cervical squamous metaplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 30 (32) | 28 (30)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Propionate/Salmeterol Combination (FSC) (N=5834) | Fluticasone Propionate (FP) (N=5845)
Asthma (Respiratory, thoracic and mediastinal disorders) | 46 | 75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.